CLINICAL TRIAL: NCT04116892
Title: Prospective, Consecutive, Non-randomized,Interventional Trial of Comparative Analysis of Large Macular Hole Surgeries
Brief Title: Comparative Analysis of Large Macular Hole Surgeries
Acronym: CAOLMHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IR001094; 2019-142 (Other: 2nd Affiliated Hospital, School of Medicine, Zhejiang University)
Record Dates: First submitted 2019-09-29; First posted 2019-10-07 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Macular Holes
Keywords: Inverted Internal Limiting Membrane Flap Technique; Large Macular Hole; Macular hole surgery
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the peeling group (Active Comparator): the internal limiting membrane was discarded
  Interventions: Procedure: the peeling group
- the Cover group (Experimental): the internal limiting membrane was peeled centripetally all the way up to the MH rim and the hinged ILM flap folded upside-down on top of the MH in order to bridge the entire retinal defect with a single layer.
  Interventions: Procedure: the Cover group
- the Fill group (Experimental): the internal limiting membrane was folded in multiple layers and deliberately "stuffed" or "packed" within the MH defect using a forceps.
  Interventions: Procedure: the Fill group

INTERVENTIONS:
Procedure: the Cover group — The internal limiting membrane around the MH was left to cover the hole
  Arms: the Cover group
Procedure: the Fill group — The internal limiting membrane around the MH was left to fill the hole
  Arms: the Fill group
Procedure: the peeling group — the internal limiting membrane was discarded
  Arms: the peeling group

SUMMARY:
This study compares the anatomical and visual outcomes in a large series of patients affected by idiopathic macular holes larger than 400 µm treated using pars plana vitrectomy and gas tamponade combined with internal limiting membrane (ILM) peeling or the inverted internal limiting membrane flap technique. A part of the participants will receive internal limiting membrane peeling,whil the other will receive the inverted internal limiting membrane flap technique.

DETAILED DESCRIPTION:
Vitrectomy is the standard treatment for idiopathic macular holes (IMHs) and is combined with removal of the internal limiting membrane (ILM) to improve anatomical outcomes.However, surgical closure is not achieved after a single operation in all cases, and patients with long-standing MHs or highly myopic eyes are challenging to treat.Various surgical strategies have been introduced to improve postoperative outcomes for these cases. Michalewska et al. have reported an inverted ILM flap technique for large MHs. The ILM around the MH was left to cover or fill the hole and showed a better anatomical closure rate and visual outcome than ILM peeling for large MHs. Nevertheless, the functional and anatomic outcomes of the ILM flap technique have not been investigated as extensively as the ILM peeling technique and have yet to be confirmed by research comparing the ILM flap technique with the conventional procedure.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic MHs, a minimum hole diameter of ≥ 400 μm, and follow-up for at least 3 months after vitrectomy.

Exclusion Criteria:

* High myopia (≥6 diopters,AL≥26.5mm), increased intraocular pressure (IOP, >21 mm Hg) or glaucoma, severe cataract, severe systemic conditions that prevent surgery, and history of ocular trauma, intraocular inflammation, retinal vascular disease, or previous ocular surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
MH status | at 3 months after surgery
  MH status (open, flat open or closed)
IS/OS line interruption width | at 3 months after surgery
  IS/OS line interruption width were gauged with spectral-domain optical coherence tomography
Change from Baseline IS/OS line interruption width at 3 months | at 3 months after surgery
  IS/OS line interruption width were gauged with spectral-domain optical coherence tomography
Baseline best-corrected visual acuity | at 3 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
Change from Baseline best-corrected visual acuity at 3 months | at 3 months after surgery
  best-corrected visual acuity were gauged with EDTRS charts,recorded in decimals and was converted to logarithm of the minimum angle of resolution units for statistical analysis
visual function | at 3 months after surgery
  visual function were gauged with national eye institute visual function questionnaire-25((NEI VFQ-25)
Change from Baseline visual function at 3 months | at 3 months after surgery
  visual function were gauged with national eye institute visual function questionnaire-25((NEI VFQ-25)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Ophthalmology, The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No